CLINICAL TRIAL: NCT03993405
Title: Cut-off Values and Adjustments for Diagnosing Sarcopenia
Brief Title: Cut-off Values of Muscle Thickness Ratio for Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ozden Ozkal, Principal Investigator, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: GO 18/506-39
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-06

CONDITIONS: Sarcopenia
Keywords: older people; muscle; ultrasound
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group:young (Active Comparator): Sixty older subjects will be evaluated in this study.
  Interventions: Other: Ultrasonographic evaluation
- Control Group:Middle-aged (Active Comparator): Sixty middle-aged subjects will be evaluated in this study.
  Interventions: Other: Ultrasonographic evaluation
- Experimental group:older (Experimental): Sixty older subjects will be evaluated in this study.
  Interventions: Other: Ultrasonographic evaluation

INTERVENTIONS:
Other: Ultrasonographic evaluation — Ultrasonographic measurement is assessment method to diagnosis of sarcopenia

SUMMARY:
The loss of muscle mass is one of the major diagnostic criteria for sarcopenia. Many methods are also used for the definition of sarcopenia. However there is no information about cut-off values in this respect in the literature. Therefore, the aim of this study is to determine the cut-off values of this ratio for confirming the diagnosis of sarcopenia.

DETAILED DESCRIPTION:
Decreases in total skeletal muscle mass are accepted to be necessary for confirming the diagnosis of sarcopenia. Many methods are also used for the definition of sarcopenia.

However, ultrasound measurements has a high sensitivity and specify for confirming the diagnosis of sarcopenia. However there is no information about cut-off values in this respect in the literature. Therefore, the aim of this study is to determine the cut-off values of this ratio for confirming the diagnosis of sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* To be a volunteer to participate
* To be an aged 18-90 years old.

Exclusion Criteria:

* Walking with assist device
* Having a visual deficits
* Having an undergone orthopedic surgery
* Having a cardiac pacemaker
* Having a hypothyroidism, diabetes mellitus, renal/hepatic failure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
Muscle thickness | 30 minutes
  Muscle thickness in millimeters by Ultrasound.
Skeletal muscle mass | 2 minutes
  Skeletal muscle mass will be evaluated by bioelectrical impedance analysis.The unit of measure is kg.

SECONDARY OUTCOMES:
Muscle strength | 15 minutes
  Muscle strength will be evaluated using an isokinetic dynamometer (Biodex Medical Systems, New York, USA). Knee and ankle muscle strength( flexion, extension, dorsiflexion and plantarflexion) will be evaluated. The unit of measure is Nm/kg.
Peripheral strength | 1 minutes
  The peripheral (handgrip) strength will be measured with a dynamometer (JAMAR).Three measurements will be taken, whose average of the three measurements will be collected. The unit of measure is kg.
Physical function | 5 minutes
  Physical function will be evaluated by short physical performance scale. The score of this scale range from 0 (worst performance) to 12 (best performance).
Anthropometric assessments | 5 minutes
  Participants waist, hip and calf circumferences will be measured by tape measure. The unit of measure is centimeters.
Balance | 1 minute
  Timed up and go test evaluates dynamic balance of participants. The timed up and go test measures the time that a patient needs to stand up from a chair, walk a 3-m distance, come back and sit back on the chair.Timed up and go test measure is second. The lower values indicates the better balance.
Body mass index | 1 minute
  Participants' weight and height will be evaluated by electronic weighing and tape measure, respectively. body mass index will be expressed in in kg/ m²

CONTACTS AND LOCATIONS:
Locations (1):
- Ozden Ozkal, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No